CLINICAL TRIAL: NCT05626907
Title: Assessing the Effect of Diet on Hypothalamic Gliosis in Humans
Brief Title: Does What You Eat Affect Your Brain
Acronym: WYE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ellen Schur, MD, MS, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY00015328; 1R01DK133356-01 (NIH)
Record Dates: First submitted 2022-09-23; First posted 2022-11-25 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Gliosis; Obesity; Eating
MeSH Terms: conditions — Gliosis; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Assigned Diet #1 (Experimental)
  Interventions: Other: Diet modification #1
- Assigned Diet #2 (Experimental)
  Interventions: Other: Diet modification #2
- Assigned Diet #3 (Other)
  Interventions: Other: Diet modification #3

INTERVENTIONS:
Other: Diet modification #1 — Participants will be provided all meals for a 14-day period. For 7 of the days, meals will be 130% of estimated daily caloric needs and for the other 7 days, meals will be low in calories, consistent with recommendations for weight loss.
  Arms: Assigned Diet #1
Other: Diet modification #2 — Participants will be provided all meals for a 14-day period. For 7 of the days, meals will be 150% of estimated daily caloric needs and for the other 7 days, meals will be meals will be low in calories, consistent with recommendations for weight loss.
  Arms: Assigned Diet #2
Other: Diet modification #3 — Participants will be provided all meals for a 14-day period to be approximately 100% of estimated daily caloric needs.
  Arms: Assigned Diet #3

SUMMARY:
The purpose of this study is to use magnetic resonance imaging (MRI) to evaluate the human hypothalamus for signs of inflammation in response to specific diets. This research may lead to a better understanding of how poor nutritional quality may lead to obesity through effects on regions of the brain known to regulate body weight.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-40 years
* Overweight: BMI 25-29.9 kg/m2
* Willing to undergo randomly assigned 14-day diet modification

Exclusion Criteria:

* History of bariatric surgery or active participation in weight-loss program
* Major medical or neurological disorder (e.g., diabetes, multiple sclerosis)
* Anemia or impaired kidney or liver function
* Known gallbladder disease or gallstones
* Hypertriglyceridemia (>350 mg/dl)
* Current use of orlistat or other weight-loss medications or other medications known to alter appetite (e.g., atypical anti-psychotics)
* More than moderate level of physical activity (>1000 met-min/wk)
* Pregnancy, menopause, or breastfeeding
* MRI contraindication (e.g., implanted metal, claustrophobia)
* Lifetime eating disorder
* Current smoking or heavy alcohol use (≥ 2 drinks per day for females and ≥ 3 drinks per day for males)
* Weight > 350 pounds (MRI limit)
* Dietary restrictions (e.g., vegan) incompatible with controlled diets

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Hypothalamic Gliosis | 7 days of diet intervention
  T2 relaxation time as measured by brain MRI

CONTACTS AND LOCATIONS:
Overall Officials: Ellen A Schur, MD, MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No